CLINICAL TRIAL: NCT04976647
Title: A Randomized, Open-Label, Multicenter, Phase II Study of HLX07 (Anti-EGFR Antibody) +HLX10 (Anti-PD-1 Antibody) With or Without Chemotherapy Versus HLX10 With Chemotherapy in First Line sqNSCLC
Brief Title: A Study of HLX07 + HLX10 With or Without Chemotherapy Versus HLX10 With Chemotherapy in First Line sqNSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX10HLX07-sqNSCLC-201
Record Dates: First submitted 2021-07-20; First posted 2021-07-26 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Squamous Non-small-cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A arm: HLX10+chemo (Active Comparator): Participants receive 300mg HLX10 IV every 3 weeks (Q3W) in combination with carboplaitin (AUC5 or 6) IV Q3W and nab-paclitaxel (260mg/m2) IV Q3W for 4-6 circle.
  Interventions: Drug: HLX10+chemo
- B arm: HLX10+HLX07+chemo (Experimental): Participants receive 300mg HLX10 IV Q3W plus 1500mg HLX07 IV Q3W with chemo.
  Interventions: Drug: HLX10+HLX07+chemo
- C arm: HLX10+HLX07 (Experimental): Participants receive 300mg HLX10 IV Q3W plus 1500mg HLX07 IV Q3W.
  Interventions: Drug: HLX10+HLX07

INTERVENTIONS:
Drug: HLX10+chemo — HLX10 300mg IV Q3W; carboplaitin (AUC5 or 6) IV Q3W + nab-paclitaxel (260mg/m2) IV Q3W for 4-6 circle
  Arms: A arm: HLX10+chemo
Drug: HLX10+HLX07+chemo — HLX07 1500mg IV q3w; HLX10 300mg IV Q3W; carboplaitin (AUC5 or 6) IV Q3W + nab-paclitaxel (260mg/m2) IV Q3W for 4-6 circle
  Arms: B arm: HLX10+HLX07+chemo
Drug: HLX10+HLX07 — HLX07 1500mg IV q3w; HLX10 300mg IV Q3W;
  Arms: C arm: HLX10+HLX07

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of HLX07 In Combination with HLX10 with or without Chemotherapy versus HLX10 with Chemotherapy in First Line Recurrent or Metastatic Squamous Non-Small Cell Lung Cancer.This study consists of three periods, screening period (28 days), treatment period and follow-up period (including safety follow-up, survival follow-up).Subjects can be enrolled into this study only if they meet inclusion criteria and do not meet exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of previously untreated, Recurrent or Metastatic Squamous Non-Small Cell Lung Cancer
* EGFR immunohistochemistry (IHC) H score ≥200 assessed by central lab
* Has measurable disease as defined by RECIST 1.1 as determined by the IRRC
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Has a life expectancy of greater than 12 weeks
* Has adequate organ function

Exclusion Criteria:

* Histologically non-squamous NSCLC must be exclused. For non-small-cell histology, if has squamous components be allowed
* Has history of such as PD-1/PD-L1、EGFR、 CTLA4 targeted therapy
* EGFR sensitivity mutation or ALK or ROS1 gene rearrangement need to be excluded
* Has had other active malignancies within 5 years or at the same time
* Has uncontrolled pleural effusion、pericardial effusion or ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 assessed by IRRC | Up to 5 years
  ORR is defined as the percentage of participants who have a Complete Response ([CR], disappearance of all evidence of disease) or Partial Response ([PR], regression of measurable disease and no new sites) per RECIST 1.1 as assessed by IRRC. ORR will be determined for each treatment arm.
Progression Free Survival (PFS) per RECIST 1.1 assessed by IRRC(Independent Radiology Review Committee) | Up to 5 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by IRRC or death due to any cause, whichever occurs first. PFS will be determined for each treatment arm

SECONDARY OUTCOMES:
Adverse Events (AE) | Up to 5 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experience an AE will be reported for each treatment arm.
Duration of Response (DOR) per RECIST 1.1 assessed by IRRC | Up to 5 years
  For participants who demonstrate CR or PR, DOR is defined as the time from first response (CR or PR) to subsequent disease progression or death from any cause, whichever occurs first. DOR will be determined for each treatment arm
Overall Survival (OS) | Up to 5 years
  OS is defined as the time from randomization to death due to any cause. OS will be determined for each treatment arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China